CLINICAL TRIAL: NCT06338046
Title: Evaluation of the Efficacy and Safety of a Shiitake Mushroom Oil-Soluble Extract (SMosE) on Skin Barrier Function, Sebum Regulation, and Adaptive Responses: Preclinical and Clinical Investigation
Brief Title: SMosE Safety and Efficacy Evaluation as a Skin Adaptogen
Acronym: SMosE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Ritamaria Di Lorenzo, PhD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EAShi23M01
Record Dates: First submitted 2024-03-23; First posted 2024-03-29 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2024-03

CONDITIONS: Sebum Production; Acne Scars; Skin Barrier to Water Loss

STUDY DESIGN:
Intervention Model Description: 2 parallel arm, double blind, randomized, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: neither the patient nor the investigator knows who is getting which treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sample A - Active treatment (Active Comparator): 28-day-treatment, with twice daily application (morning and evening) of a cosmetic formula containing NC65 - Vita D-Light at 0.5 %w/w. The cosmetic formula is a w/o emulsion done with cosmetic-grade ingredients according to GMP. The designed quantity to be applied on the face is approximately 2 mg.
  Interventions: Other: Corthellus Shiitake(Mushroom) Extract
- Sample B - Placebo treatment (Placebo Comparator): 28-day-treatment, with twice daily application (morning and evening) of a cosmetic formula containing the same ingredient of the active treatment except for NC65 - Vita D-Light at 0.5 %w/w. The cosmetic formula is a w/o emulsion done with cosmetic-grade ingredients according to GMP. The designed quantity to be applied on the face is approximately 2 mg.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Corthellus Shiitake(Mushroom) Extract — topical treatment with Corthellus Shiitake(Mushroom) Extract
  Other Names: NC65 - Vita D-Light
  Arms: Sample A - Active treatment
Other: Placebo — topical treatment with a placebo cosmetic formula
  Other Names: Sample B
  Arms: Sample B - Placebo treatment

SUMMARY:
This study evaluates the biological activity, safety, and clinical efficacy of SMosE (Shiitake Mushroom Oil-Soluble Extract), a topical cosmetic ingredient developed to support skin barrier function, adaptogenic responses, and sebum balance.

The investigation integrates preclinical in vitro studies, ex vivo human skin explant experiments, and a randomized, double-blind, placebo-controlled clinical trial. Preclinical models were used to explore the molecular mechanisms of action of SMosE on epidermal differentiation and barrier-related markers. The clinical phase assessed the effects of a topical formulation containing SMosE on skin hydration, transepidermal water loss, sebum production, and skin surface features in adult volunteers.

DETAILED DESCRIPTION:
Background and Rationale:

Skin homeostasis depends on the integrity of the epidermal barrier, balanced sebum production, and the ability of the skin to adapt to environmental stressors. Cosmetic ingredients with adaptogenic properties are increasingly investigated as non-invasive strategies to support these functions.

SMosE is an oil-soluble extract obtained from Lentinus edodes (shiitake mushroom), developed for topical use. Preliminary data suggest that SMosE may promote epidermal differentiation, improve barrier-related protein expression, and modulate sebum-related pathways.

Preclinical Evaluation:

Ex Vivo Human Skin Explant Study:

To confirm biological relevance in intact human tissue, ex vivo studies were performed on human skin explants. Human skin explants were obtained from three healthy female donors, aged 26 to 40 years, who underwent abdominoplasty or breast reduction surgery. All donors provided written informed consent for the use of their skin tissues in accordance with the Declaration of Helsinki. Then, protein expression of epidermal differentiation and barrier markers, including cytokeratin 10 and claudin-1, was evaluated by immunofluorescence microscopy.

Clinical Study Design:

The clinical phase was designed as a randomized, double-blind, placebo-controlled, parallel-group cosmetic study conducted at a single center.

A total of 40 adult male and female volunteers with oily and/or acne-prone skin were enrolled and randomized in a 1:1 ratio to receive either: a topical formulation containing SMosE, or a placebo formulation identical in composition except for the absence of the active ingredient. Participants applied the assigned product to the face once daily for 28 consecutive days.

Clinical Assessments:

Skin evaluations were performed at baseline and during follow-up visits under controlled environmental conditions using validated, non-invasive instruments to assess hydration, barrier function, sebum production, and skin surface features.

Safety and Ethics :

Skin tolerability was assessed prior to and throughout the study. Adverse events were monitored and recorded. All participants provided written informed consent. The study was conducted in accordance with the principles of the Declaration of Helsinki and applicable guidelines for cosmetic clinical research.

ELIGIBILITY:
Inclusion Criteria:

* Subjects scheduled for eligibility screening at the study site
* Female or Male sex
* Subjects with acne prone skin or skin with scar from acne
* Subjects exposed to sunlight for at least 4 hours a day
* Signing the informed consent form written by the investigators
* Certifying not taking part in another clinical study that could interfere with the current one
* Affirming the truth of the personal information declared to the technical staff
* Capable of following directions and reliable to respect the constraints of the protocol
* Free to ensure the visits to the Research Lab
* Subjects with self-perceived
* Subjects may have mild to sensitive and stressed skin

Exclusion Criteria:

* Female subjects who are pregnant, breastfeeding, or planning a pregnancy
* Subjects with severe overall photodamage as determined by the Investigator.
* Subjects who have any dermatological disorder, which in the investigator's opinion, may interfere with the accurate evaluation of the subject's skin, including rosacea, acne, and excessively oily or dry skin.
* Subjects who have demonstrated a previous hypersensitivity reaction to any of the ingredients of the study products.
* Subjects' use of any medications that are known to potentially cause changes in the facial skin as determined by the Investigator.
* Subjects who spend excessive time out in the sun.
* Subjects who are unwilling or unable to comply with the requirements of the protocol.
* Subjects deprived of freedom by administrative or legal decision or under guardianship
* Subjects planning hospitalization during the study
* Subjectsaving received vaccination within 2 weeks before the study or intending to be vaccinated during the study
* Subjects with diseases in the period immediately preceding the current study under treatment topically or systemically with any drug that may affect the outcome of the test, particularly: systemic retinoids within 6 months, topical retinoids within 2 months anti-inflammatory or antihistamine products within the 2 weeks antibiotics within 2 weeks medication for malignancy (of any kind) within 5 years desensitization treatment within 6 months
* Subjects in treatments with topical products based on alpha and beta-hydroxy acids in the 45 days before the start of the study
* Subjects reactive to sun/having photosensitivity.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Soothing Test | 2 months
  SOOTHING ACTION EFFICACY

SECONDARY OUTCOMES:
Detox and adaptogen Test | 8 months
  SKIN ADAPTOGEN AND SEBUM BALANCE EFFICACY

CONTACTS AND LOCATIONS:
Overall Officials: Ritamaria Di Lorenzo, Principal Investigator — Federico II University
Locations (1):
- RD Cosmetics Lab - Pharmacy Department, University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: No